CLINICAL TRIAL: NCT05229146
Title: Reducing Maternal Delay Discounting as a Target Mechanism to Decrease Harsh Parenting and Improve Child Mental Health Outcomes in a Traditionally Underserved Community
Brief Title: Improving Future Thinking Among Mothers to Reduce Harsh Parenting and Improve Child Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Maryland, College Park (Other); University of Kansas (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Julia Felton, Assistant Scientist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NHP: 15407-31
Record Dates: First submitted 2022-01-18; First posted 2022-02-08 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Behavioral Health
Keywords: episodic future thinking; delay discounting; parent-child relations; low income; substance use treatment; peer recovery coach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Episodic Future Thinking (Experimental): Mothers will receive episodic future thinking (EFT). Mothers will meet with a "peer mother" who will administer the EFT intervention, including generation of several specific future events reflecting positive interactions with their child. We will also teach each parent a behavioral parent training element called Special Play Time. Following this session, mothers will receive daily text messages over the course of two weeks including a reminder cue generated as part of the EFT and a prompt to remember these episodes in vivid detail.
  Interventions: Behavioral: Episodic Future Thinking

INTERVENTIONS:
Behavioral: Episodic Future Thinking — Episodic future thinking (EFT) includes a focus on generating detailed and vivid descriptions of future events. For the current intervention, EFT will be modified to have mothers describe specific events with their children.

SUMMARY:
Parents of children from impoverished communities are disproportionately more likely to engage in harsh physical discipline, which can lead to serious clinical outcomes, including suicidal ideation and attempts. One mechanism linking low resource environments and maladaptive parenting strategies is maternal delay discounting, or the tendency to value smaller, immediate rewards (such as stopping children's misbehavior via physical means) relative to larger, but delayed rewards (like improving the parent-child relationship). This study will examine the efficacy of implementing a low-cost, brief intervention targeting the reduction of maternal delay discounting to inform broader public health efforts aimed at improving adolescent mental health outcomes in traditionally underserved communities.

DETAILED DESCRIPTION:
Harsh parenting is associated with serious and costly mental health problems among youth, including substance use, mood disorders, and suicidal ideation and behaviors. Of concern, these parenting practices are most common among families from impoverished communities; however, many behaviorally-based parenting interventions do not take into account the unique mechanisms linking environmental disadvantage to parenting approaches. While the causes of harsh parenting are complex and varied, one such mechanism may be parents' tendencies to prioritize immediate rewards (such as stopping a child's misbehavior via physical punishment like spanking and hitting) relative to larger, but delayed rewards (including improved parent-child relationship quality), known as delay discounting. This case series will examine the efficacy of episodic future thinking (EFT) to target reduction of parenting-related delay discounting. Outcomes will evaluate the effect of EFT on reducing maternal delay discounting and harsh parenting, and improving child clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Be the mother from the Flint area of a child between the ages of 5-10 who can provide legal consent for that child to participate in this study
2. Self-report that the child lives with them for at least 50% of the time
3. Willing to participate in the study
4. Able to participate in written assessments and an intervention conducted in English
5. Have a working cell phone that can receive and send text messages and be willing to receive/send text messages as part of the study
6. Have a phone or device that's able to use video conferencing software

Exclusion Criteria:

1. Self-disclosed active suicidality/homicidality
2. Self-disclosed current bipolar disorder, schizophrenia, or psychosis
3. Current and ongoing involvement with child protective services

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RL Jones Community Outreach Center, Flint, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 mothers of children ages 5-10 provided informed consent for themselves and (n=24) their children.
Period: Overall Study
Arm/Group | Episodic Future Thinking
Started (Completed baseline assessment battery.) | 48 (24 mothers (out of the 24 mothers that consented) completed baseline measures including providing data on n=24 children.)
Completed Intervention With Peer Mother. | 34 (17 mothers (out of the 24 mothers that consented) completed the intervention with a peer mother; and 17 children.)
Completed (Completed the two-week post-intervention assessment battery.) | 32 (16 mothers (out of the 24 mothers that consented) completed the two-week follow-up intervention; and n=16 children.)
Not Completed | 16

BASELINE CHARACTERISTICS:
Population: 24 dyads (24 mothers of children 5-10 and reported on their n=24 children). Mothers reported demographic data for themselves and their children.
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants] — Population: Age data on mothers in sample.
  Participants
    Mothers: number analyzed (Participants) | 24
    Mothers: <=18 years | 0
    Mothers: Between 18 and 65 years | 24
    Mothers: >=65 years | 0
    Children: number analyzed (Participants) | 24
    Children: <=18 years | 24
    Children: Between 18 and 65 years | 0
    Children: >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Continuous age data is reported separately for mothers and their children.
  years
    Mothers: number analyzed (Participants) | 24
    Mothers | 35.5 (6.1)
    Children: number analyzed (Participants) | 24
    Children | 7.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data is reported separately for mothers and children.
  Participants
    Mothers: number analyzed (Participants) | 24
    Mothers: Female | 24
    Mothers: Male | 0
    Children: number analyzed (Participants) | 24
    Children: Female | 10
    Children: Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data is reported for mothers and children separately.
  Participants
    Mothers: number analyzed (Participants) | 24
    Mothers: Hispanic or Latino | 0
    Mothers: Not Hispanic or Latino | 24
    Mothers: Unknown or Not Reported | 0
    Children: number analyzed (Participants) | 24
    Children: Hispanic or Latino | 1
    Children: Not Hispanic or Latino | 23
    Children: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data is reported for mothers and children separately.
  Participants
    Mothers: number analyzed (Participants) | 24
    Mothers: American Indian or Alaska Native | 1
    Mothers: Asian | 0
    Mothers: Native Hawaiian or Other Pacific Islander | 0
    Mothers: Black or African American | 8
    Mothers: White | 15
    Mothers: More than one race | 0
    Mothers: Unknown or Not Reported | 0
    Children: number analyzed (Participants) | 24
    Children: American Indian or Alaska Native | 1
    Children: Asian | 0
    Children: Native Hawaiian or Other Pacific Islander | 0
    Children: Black or African American | 8
    Children: White | 15
    Children: More than one race | 0
    Children: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Monetary Choice Questionnaire
Description: The brief Monetary Choice Questionnaire (MCQ) is a 21-item binary-choice task that asks participants to select between two hypothetical monetary amounts: a smaller reward available immediately (e.g. $49 today) or a larger reward available after a delay (e.g. $60 in 89 days). "Larger later" amounts are separated into small, medium and large magnitudes. For the purposes of this study, to limit participant burden, we administered only small and large magnitude subscales, resulting in a total number of 14 items. The measure is scored to derive a single "total score" discounting rate k, with larger values reflecting greater preference for smaller sooner reward. Because k distributions are typically skewed, post-hoc natural logarithmic transformations were performed, resulting in normal distributions; thus, there is no maximum and minimum value. The MCQ has been shown to have strong psychometric properties among adults and correlates with real rewards, as well as real-world risk behaviors.
Time Frame: Baseline, 1 week, 4 weeks
Population: Mothers who completed the the MCQ both at baseline and immediately following the intervention (approximately 1 week later).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 11
score on a scale
  Baseline Assessment | -3.86 (1.42)
  Immediately Post-Intervention (1 week) | -4.13 (1.19)
  Post-intervention (2 weeks after intervention, 4 weeks after baseline) | -4.33 (1.68)
Statistical Analysis 1: Comparison: Episodic Future Thinking; One-sided paired-samples t-test comparing baseline to responses immediately following the intervention (approximately one week after baseline); Test type: Superiority; p = .191, t-test, 1 sided — No adjustment for multiple comparisons; t-statistic = .913, df = 10
Statistical Analysis 2: Comparison: Episodic Future Thinking; One-sided paired-samples t-test comparing baseline to responses at two week follow-up (approximately four weeks after baseline); Test type: Superiority; p = .043, t-test, 1 sided — Not adjusted for multiple comparisons; t-statistic = 1.92, df = 9

2. Primary Outcome: Change in Consideration of Future Consequences Scale-Parenting Score
Description: The Consideration of Future Consequences Scale-Parenting Adapted (CFCS-14-PA) is a 14-item self-report questionnaire composed of two subscales reflecting either immediate or future orientation related to parents interactions with their children. Items range from "not at all like me" (1) to "very much like me" (5) and are summed to create future or immediate orientation subscale, each composed of 7 items with score ranges from 7-35. Lower scores on the future orientation and higher scores on the immediate orientation subscales are associated with less future orientation and predictive of less engagement in health behaviors. The measure has been used extensively among adult samples and demonstrates strong reliability and validity. Change in CFCS-14-PA score is measured by comparing scores at the post-intervention assessment (approximately 4 weeks after baseline) with baseline scores.
Time Frame: Baseline, 4 weeks
Population: All mothers (participants) that completed this measure at baseline assessment (one participant did not complete this measure).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 23
score on a scale
  Baseline Future Orientation Subscale | 29.7 (4.5)
  Baseline Immediate Orientation Subscale | 15.7 (4.5)
  Follow-up Future Orientation Subscale | 31.3 (2.7)
  Follow-up Immediate Orientation Subscale | 16.3 (3.5)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Comparison is between future orientation subscale pre- and post-subscale scores; Test type: Superiority; p = .319, t-test, 2 sided — No adjustments were made. DF = 15; Mean Difference (Final Values) = -1.03
Statistical Analysis 2: Comparison: Episodic Future Thinking; Comparison between immediate-orientation subscales; Test type: Superiority; p = .488, t-test, 2 sided; No adjustments were made. DF = 15; Mean Difference (Final Values) = -.711

3. Secondary Outcome: Change in Dyadic Parent-Child Interaction Coding System Scores
Description: Parents and their children will complete a 20-minute interaction task, including 5 min. of free play, a 10 min. "homework" task, and a 5 min. clean up task. Wualitvey of parent-childre interactions were coded using the Dyadic Parent-Child Interaction Coding System (DPICS). The task has 7 subscales, yielding 2 composite scores: positive parenting (a sum of: unlabeled praise, labeled praise, positive touch, reflection, and behavior description) and negative parenting (a sum of: negative talk and negative touch). Each instance of a behaviors described in the subscale (e.g., a parent giving unlabeled praise) is coded as one "point" and summed into a subscale (no max or min values). Higher values indicate greater positive or negative parenting. A score is given to the dyad (not individuals scores for parent/child). Change in parenting is calculated by comparing baseline scores with scores at the post-intervention sessions (approximately 4 weeks after baseline).
Time Frame: Baseline, 4 weeks
Population: 11 dyads , including mothers (n=11) and their children (n=11), participated in the parent child interaction task at both the pre-intervention and post-intervention assessment. Please note that scores are given at the dyadic level (in other words, there is a single score for each dyad).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 11
score on a scale
  Positive Parenting Composite Score Pre-Intervention | 10.73 (7.96)
  Positive Parenting Composite Score Post-Intervention | 9.91 (8.68)
  Negative Parenting Composite Score Pre-Intervention | 8.82 (7.48)
  Negative Parenting Composite Score Post-Intervention | 9.18 (6.55)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Performed a paired-samples one-sided t-test comparing positive parenting before the intervention to after the intervention; Test type: Superiority; p = .34, t-test, 1 sided; No adjustments were made. DF = 10; Mean Difference (Final Values) = .438
Statistical Analysis 2: Comparison: Episodic Future Thinking; Performed a one-sided paired-samples t-test to compare negative parenting before and after the intervention; Test type: Superiority; p = .362, t-test, 1 sided; No adjustments were made. DF = 10; Mean Difference (Final Values) = -.363

4. Secondary Outcome: Change in Alabama Parenting Questionnaire Score
Description: The Alabama Parenting Questionnaire (APQ) is a 42-item self-report measure of parenting behaviors which yields five subscales: (1) positive involvement with children (range 10-50, higher = more involvement), (2) use of positive parenting strategies (range 6-30, higher = more positive strategies), (3) poor parental monitoring/supervision (range 10-50, higher = worse supervision), (4) inconsistent discipline (range 6-30, higher = more inconsistent discipline), and (5) use of corporal punishment (higher = more corporal punishment). Items are summed to create subscale scores. Change in each of the five APQ subscale scores will be measured by comparing post-intervention scores (approximately 4 weeks after baseline) with baseline scores.
Time Frame: Baseline, 4 weeks
Population: Mothers who completed the APQ measure at baseline and at follow-up (approximately four weeks later).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 16
score on a scale
  Involvement Subscale Pre-Intervention | 40.13 (4.47)
  Involvement Subscale Post-intervention | 43 (4.93)
  Positive Parenting Subscale Pre-Intervention | 25.89 (3.55)
  Positive Parenting Subscale Post-Intervention | 26.50 (2.99)
  Inconsistent Parenting Subscale Pre-Intervention | 15.44 (3.68)
  Inconsistent Parenting Subscale Post-Intervention | 13.59 (4.25)
  Corporal Punishment Subscale Pre-Intervention | 5.94 (2.05)
  Corporal Punishment Subscale Post-Intervention | 5.00 (1.86)
  Poor parental monitoring Subscale Pre-Intervention | 12.81 (2.64)
  Poor parental monitoring Subscale Post-Intervention | 11.72 (2.22)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Used a one-sided paired samples t-test to examine changes in the parental involvement subscale from pre-intervention to post-intervention (approximately 4 weeks later); Test type: Superiority; p < .001, t-test, 1 sided; No adjustments, DF = 15; Mean Difference (Final Values) = -3.77
Statistical Analysis 2: Comparison: Episodic Future Thinking; Used a one-sided paired samples t-test to examine changes in the positive parenting subscale from pre-intervention to post-intervention (approximately 4 weeks later); Test type: Superiority; p = .137, t-test, 1 sided; Median Difference (Final Values) = -1.14
Statistical Analysis 3: Comparison: Episodic Future Thinking; Used a one-sided paired samples t-test to examine changes in the inconsistent discipline subscale from pre-intervention to post-intervention (approximately 4 weeks later); Test type: Superiority; p = .018, t-test, 1 sided; No adjustments; DF = 15; Mean Difference (Final Values) = 2.31
Statistical Analysis 4: Comparison: Episodic Future Thinking; Used a one-sided paired samples t-test to examine changes in the use of corporal punishment subscale from pre-intervention to post-intervention (approximately 4 weeks later); Test type: Superiority; p = .015, t-test, 1 sided; No adjustments; DF = 15; Mean Difference (Final Values) = 2.39
Statistical Analysis 5: Comparison: Episodic Future Thinking; Used a one-sided paired samples t-test to examine changes in the poor parental monitoring/supervision subscale from pre-intervention to post-intervention (approximately 4 weeks later); Test type: Superiority; p = .021, t-test, 1 sided; Mean Difference (Final Values) = 2.23

5. Secondary Outcome: Change in Emotion Regulation Checklist
Description: Parents will report on children's emotion regulation using the Emotion Regulation Checklist (ERC). Items are rated from 1 to 4 and summed to create subscales. The ECR includes 24 items. 23 items are used in computing two subscales: (1) emotion regulation (range 8 to 32, higher = greater emotion regulation) and (2) lability/negativity (range 15 to 60, higher = greater lability/negativity); the 24th item does not load onto either subscale and is not used in the current analyses. The measure is widely used and validated for parent-report of older children and young adolescents.
Time Frame: Baseline, 4 weeks
Population: Mothers who completed Emotion Regulation Checklist and pre- and post-intervention (approximately 4 weeks later).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 16
score on a scale
  Emotion Regulation Subscale Pre-Intervention | 25.63 (3.61)
  Emotion Regulation Subscale Post-Intervention | 25.00 (3.06)
  Lability/Negativity Subscale Pre-Intervention | 30.13 (8.88)
  Lability/Negativity Subscale Post-Intervention | 29.00 (6.58)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Used a one-sided paired-samples t-test to examine changes in emotion regulation subscale from pre-intervention to post-intervention; Test type: Superiority; p = .197, t-test, 1 sided; No adjustments; DF = 15; Mean Difference (Final Values) = .878
Statistical Analysis 2: Comparison: Episodic Future Thinking; Used a one-sided paired-samples t-test to examine changes in lability/negativity subscale from pre-intervention to post-intervention; Test type: Superiority; p = .203, t-test, 1 sided; No adjustments, DF = 15; Mean Difference (Final Values) = .857

6. Secondary Outcome: Client Satisfaction Questionnaire
Description: Following the completion of the intervention, mothers will complete the Client Satisfaction Questionnaire (CSQ), which evaluates participant satisfaction with the intervention. Nine items are ranked from 1 to 4 and summed to create a total score (range 9-36, higher = greater satisfaction). The measure is used across a number of intervention studies and has been shown to be reliable and valid in adult samples.
Time Frame: 4 weeks
Population: Participants who completed the CSQ measure at follow-up (approximately 4 weeks after the intervention).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 15
score on a scale | 29.73 (5.38)

ADVERSE EVENTS:
Time Frame: Participants were involved in the study for approximately four weeks. Thus, four weeks is the period of time used below.
Arm/Group | Episodic Future Thinking
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT05229146/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT05229146/SAP_001.pdf